CLINICAL TRIAL: NCT05938465
Title: A Phase 1b/2 Study to Demonstrate the Safety and Efficacy of EXE-346 Live Biotherapeutic to Reduce High Bowel Movement Frequency in Subjects With an Ileal Pouch-Anal Anastomosis (PROF). The "PROF" Study.
Brief Title: Study of EXE-346 Live Biotherapeutic to Reduce High Bowel Movement Frequency in Subjects With an IPAA (PROF)
Acronym: PROF
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Exegi Pharma, LLC (Industry)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28193
Record Dates: First submitted 2023-05-30; First posted 2023-07-10 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Ileal Pouch
Keywords: Pouchitis; Pouch; Ileal Pouch Anastomosis; IPAA
MeSH Terms: conditions — Pouchitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase 1b Open Label (Experimental): EXE-346 live biotherapeutic product, 1500x10^9 colony forming units (CFU) twice daily (BID), 4 weeks
  Interventions: Biological: EXE-346
- Phase 2: Active Arm (Experimental): EXE-346 live biotherapeutic product, 1500x10^9 CFU BID, 8 weeks
  Interventions: Biological: EXE-346
- Phase 2: Placebo Arm (Placebo Comparator): Powder containing same inactive ingredients as EXE-346 but none of the active ingredients, BID, 8 weeks
  Interventions: Other: Placebo
- Phase 2 Open Label Extension (optional) (Experimental): EXE-346 live biotherapeutic product, 1500x10^9 CFU BID, 8 weeks
  Interventions: Biological: EXE-346

INTERVENTIONS:
Biological: EXE-346 — EXE-346 contains a proprietary, fixed-dose, lyophilized blend of 8 strains of gram positive, lactic acid bacteria. EXE-346 excipients are maltose and silicon dioxide.
  Arms: Phase 1b Open Label; Phase 2 Open Label Extension (optional); Phase 2: Active Arm
Other: Placebo — Placebo contains excipients maltose and silicon dioxide.
  Arms: Phase 2: Placebo Arm

SUMMARY:
The aim of this study is to assess the safety and preliminary efficacy of treatment with EXE-346, a live biotherapeutic, which may reduce bowel movement frequency in patients with an ileal pouch-anal anastomosis (IPAA) and lead to a higher quality of life.

DETAILED DESCRIPTION:
The aim of this study is to assess the safety and preliminary efficacy of treatment with EXE-346 which may reduce bowel movement frequency in patients with an IPAA and lead to a higher quality of life. EXE-346 is a live biotherapeutic product containing a fixed proportion mixture of 8 individual bacterial strains.

The Phase 1b part of the study is an open label (OL), single-arm study to assess the safety of EXE-346 administered orally for up to 4 weeks.

The Phase 2 part of the study is a randomized, double-blinded study to assess the safety and efficacy of the same dose of EXE-346 administered orally for up to 8 weeks, compared with placebo. Subjects who complete the Phase 2 double-blinded part of the study will be eligible to participate in an optional open label extension phase to receive EXE-346 for up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria - Phase 1b Only

1. Subject is a male or female and is between the age of 18 to 70 years, inclusive, at screening.
2. Subject has had a documented pouchoscopy within 12 months prior to screening.
3. Subject or the subject's legally authorized representative is willing and able to provide written informed consent prior to the initiation of any study-related procedures.
4. Subject has an average daily bowel movement frequency of at least 10 bowel movements recorded during screening and has correctly completed at least 7 days of eDiary entries during the screening period (Days -13 to 0).

Inclusion Criteria - Phase 2 Double-Blinded Part Only

1. Subject is a male or female and is aged 18 years or older at screening.
2. Subject is willing and able to provide written informed consent prior to the initiation of any study-related procedures.
3. Subject has an average daily bowel movement frequency of at least 10 bowel movements recorded during screening and has correctly completed at least 7 days of eDiary entries during the screening period (Days -21 to 0).

Inclusion Criteria - Both Phase 1b and Phase 2 Double-Blinded Parts

1. Subject has had an IPAA for at least 6 months prior to screening.
2. Female subjects of childbearing potential must have a negative serum pregnancy test result at screening and must not be lactating and/or breastfeeding.
3. Subjects (female subjects of childbearing potential and male subjects with partners of childbearing potential) must agree to use proper contraceptive methods (see Section 13.2 for contraceptive guidance) to avoid pregnancy during the study. Nonchildbearing potential is defined as at least 6 weeks after a hysterectomy with or without surgical bilateral oophorectomy or postmenopausal (at least 12 months since natural amenorrhea).

Inclusion Criteria - Optional Open-Label Extension Phase Only

1. Subjects must have completed the Phase 2 double-blinded part of the study and are willing to participate in the optional open-label extension phase.

   Note: Subjects who discontinued study treatment in the Phase 2 double-blinded part but who have remained in the study for safety monitoring are eligible for continued safety monitoring in the optional open-label extension phase; however, study treatment will not be re-started in such subjects.
2. Subjects must understand the study procedures, the risks involved, and are willing to continue to adhere to the study visit/protocol schedule.

Exclusion Criteria Subjects meeting any of the criteria specified below for the study phase in which they are enrolling will be excluded from the study.

Exclusion Criteria - Phase 1b Only

1. Subject has Crohn's-like disease of the pouch, as indicated by their most recent pouchoscopy during the 12 months prior to screening.
2. Subject has a stricture of the IPAA or afferent limb stricture, as indicated by their most recent pouchoscopy during the 12 months prior to screening.
3. Subject has taken biologics, azathioprine, or methotrexate within the 12 weeks prior to screening or systemic steroids within 4 weeks of screening.
4. Subject has a positive reverse transcriptase-PCR diagnostic test for SARS-CoV-2 within the 14 days prior to screening.
5. Subject has uncontrolled hypertension (systolic pressure >160 mm Hg or diastolic pressure >95 mm Hg on at least 2 measures performed at least 10 minutes apart) at screening.

Exclusion Criteria - Phase 2 Double Blinded Part Only

1. Subject has Crohn's-like disease of the pouch, as indicated by the pouchoscopy conducted during study screening.
2. Subject has isolated severe cuffitis without pouch inflammation (endoscopic mPDAI score of 2 or lower), as indicated by the pouchoscopy conducted during study screening.
3. Subject has a clinically significant stricture of the IPAA or afferent limb stricture which requires surgery or recurrent dilations more than every 3 months, as indicated by the pouchoscopy conducted during study screening. Subjects who have a planned dilation during the active study period are excluded (dilation during the screening pouchoscopy is allowed).
4. Subject has taken biologics, azathioprine, methotrexate or small molecules (e.g., JAK inhibitors, S1P receptor modulators) within the 12 weeks prior to screening or systemic steroids within 4 weeks prior to screening.
5. Subject has a positive reverse transcriptase-PCR diagnostic test for SARS-CoV-2 within the 7 days prior to screening, per subject self report.
6. Subject has an average daily bowel movement frequency of >25 bowel movements recorded during the screening period (Days -21 to 0).
7. Subject is taking opioid therapy as a long-term treatment or has taken opioids within 2 weeks prior to screening.
8. Subject has taken probiotics within 2 weeks prior to screening.
9. Subject has previously received EXE-346 for any duration. Subjects who participated in Phase 1b are excluded from Phase 2.
10. Subject has a concurrent, clinically significant, serious, unstable or uncontrolled medical or psychiatric condition that, in the opinion of the investigator, might confound study results, pose additional risk to the subject, or interfere with the subject's ability to participate fully in the study.

Exclusion Criteria - Both Phase 1b and Phase 2 Double-Blinded Part

1. Subject has enterocutaneous or recto- or pouch-vaginal fistula.
2. Subject has active Clostridium difficile infection.
3. Subject has known or suspected active CMV infection.
4. Subject initiated a new treatment with antibiotics or antimotility therapies within the 2 weeks prior to screening or plans to start a new or change doses of a current treatment during the study period (screening visit through the safety follow-up visit [Day 57 in the Phase 1b part or Day 71 in the Phase 2 part]). Subjects taking antibiotics to treat antibiotic-dependent pouchitis or antidiarrheal medication are eligible for the study provided they have been on the therapy at a stable dose for at least 2 weeks prior to screening.
5. Subject is taking NSAIDs as a long-term treatment (ie, consistent use for at least 4 days/week each month). Acute use of NSAIDs is allowed.
6. Subject has a known history or positive test during screening for HIV, HIV-1, HIV-2, or active HBV or HCV. Active HCV infection is defined as a subject with a positive hepatitis C antibody and detectable hepatitis C viral load RNA.
7. Subject has a history of malignancy within the 5 years prior to screening, with the exception of nonmelanoma skin cancer that has been treated with no evidence of recurrence, treated cervical dysplasia, or treated in situ grade 1 cervical cancer.
8. Subject has estimated glomerular filtration rate <30 mL/min/1.73 m2 at screening.
9. Subject has known hypersensitivity to EXE-346 or any product components.
10. Female subject is pregnant or lactating and/or breastfeeding.
11. Subject has participated in any clinical study of an approved or nonapproved investigational medicinal product within the 30 days prior to screening.
12. Subject has any disorder that, in the investigator's opinion, might jeopardize the subject's safety or compliance with the protocol, including but not limited to:

    1. Decompensated liver disease
    2. Elevation of AST, ALT, or bilirubin >2 × ULN
    3. Primary sclerosing cholangitis with elevated transaminases

Exclusion Criteria - Optional Open-Label Extension Phase Only

1. Subjects who have developed any medical or psychologic condition, which was excluded in the Phase 2 double-blinded part of the study or in the opinion of the investigator and/or medical monitor might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements, or to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Incidence, Severity, Relatedness, and Frequency of Treatment Emergent Adverse Events (TEAE) and Serious Adverse Events (SAE) | 4 weeks
  To assess the safety of EXE-346 using incidence, severity, relationship to study treatment, and frequency of treatment emergent adverse events (TEAE) and serious adverse events (SAE).
Phase 1b: Number of Participants with Abnormal Physical Examinations | 4 weeks
  To assess the safety of EXE-346 using abnormal findings in physical examinations after the start of study treatment that suggest a clinically significant worsening of medical issue.
Phase 1b: Number of Participants with Abnormal Vital Signs | 4 weeks
  To assess the safety of EXE-346 using abnormal findings in vital sign readings after the start of study treatment that suggest a clinically significant worsening of medical issue, including blood pressure.
Phase 1b: Number of Participants with Abnormal Safety Labs | 4 weeks
  To assess the safety of EXE-346 using markedly abnormal findings in safety labs after the start of study treatment that suggest a clinically significant worsening of medical issue.
Phase 1b: Study Treatment Discontinuation Due to Treatment Emergent Adverse Events (TEAEs) | 4 weeks
  To assess the safety of EXE-346 using study treatment discontinuation due to TEAE(s).
Phase 2: Incidence, Severity, Relatedness, and Frequency of Treatment Emergent Adverse Events (TEAE) and Serious Adverse Events (SAE) | 8 weeks
  To assess the safety of EXE-346 using incidence, severity, relationship to study treatment, and frequency of TEAEs and SAEs.
Phase 2: Number of Participants with Abnormal Physical Examinations | 8 weeks
  To assess the safety of EXE-346 using abnormal findings in physical examinations after the start of study treatment that suggest a clinically significant worsening of medical issue.
Phase 2: Number of Participants with Abnormal Vital Signs | 8 weeks
  To assess the safety of EXE-346 using abnormal findings in vital sign readings after the start of study treatment that suggest a clinically significant worsening of medical issue, including blood pressure.
Phase 2: Number of Participants with Abnormal Safety Labs | 8 weeks
  To assess the safety of EXE-346 using markedly abnormal findings in safety labs after the start of study treatment that suggest a clinically significant worsening of medical issue.
Phase 2: Study Treatment Discontinuation Due to Treatment Emergent Adverse Events (TEAEs) | 8 weeks
  To assess the safety of EXE-346 using study treatment discontinuation due to TEAE(s).
Phase 2: Change in Total Daily Bowel Movement Frequency | 8 weeks
  To assess the efficacy of EXE-346 to reduce the total daily bowel movement frequency using change in average daily bowel movement frequency from baseline to each post-baseline week
Phase 2 Open Label: Incidence, Severity, Relatedness, and Frequency of Treatment Emergent Adverse Events (TEAE) and Serious Adverse Events (SAE) | 8 weeks
  To assess the safety of EXE-346 using incidence, severity, relationship to study treatment, and frequency of TEAEs and SAEs.
Phase 2 Open Label: Number of Participants with Abnormal Physical Examinations | 8 weeks
  To assess the safety of EXE-346 using abnormal findings in physical examinations after the start of study treatment that suggest a clinically significant worsening of medical issue.
Phase 2 Open Label: Number of Participants with Abnormal Vital Signs | 8 weeks
  To assess the safety of EXE-346 using abnormal findings in vital sign readings after the start of study treatment that suggest a clinically significant worsening of medical issue, including blood pressure.
Phase 2 Open Label: Number of Participants with Abnormal Safety Labs | 8 weeks
  To assess the safety of EXE-346 using markedly abnormal findings in safety labs after the start of study treatment that suggest a clinically significant worsening of medical issue.
Phase 2 Open Label: Study Treatment Discontinuation Due to Treatment Emergent Adverse Events (TEAEs) | 8 weeks
  To assess the safety of EXE-346 using study treatment discontinuation due to TEAE(s).

SECONDARY OUTCOMES:
Phase 1b: Bowel Movement Frequency | 4 weeks
  To assess the effect of EXE-346 on bowel movement frequency using change in average daily bowel movement frequency from baseline to each post-baseline week
Phase 1b: Nighttime Awakening Frequency | 4 weeks
  To assess the effect of EXE-346 on nighttime awakening frequency using change in average nighttime awakenings for bowel movements from baseline to each post-baseline week
Phase 1b: Bowel Movement Consistency | 4 weeks
  To assess the effect of EXE-346 on bowel movement consistency using change in average consistency of daily bowel movements from baseline to each post-baseline week
Phase 2: Nighttime Awakening Frequency | 8 weeks
  To assess the effect of EXE 346 on nighttime awakening frequency using change in average nighttime awakenings for bowel movements from baseline to each post-baseline week
Phase 2: Bowel Movement Consistency | 8 weeks
  To assess the effect of EXE-346 on bowel movement consistency using change in average consistency of daily bowel movements from baseline to each post-baseline week

OTHER OUTCOMES:
Phase 1b: Change in Fecal Calprotectin Level | 4 weeks
  To evaluate the effect of EXE-346 on fecal calprotectin levels after 4 weeks. The change from baseline fecal calprotectin level will be evaluated at Day 15 and Day 29.
Phase 2: Change in mPDAI Score | 8 weeks
  To evaluate the effect of EXE-346 on the mPDAI total score from baseline to day 57.
Phase 2: Change in Clinical Subscore of mPDAI | 8 weeks
  To evaluate the effect of EXE-346 on the mPDAI clinical subscores after 8 weeks. Change from baseline clinical subscores will be calculated at Day 15, Day 29, and Day 57.
Phase 2: Change in Endoscopic Subscore of mPDAI | 8 weeks
  To evaluate the effect of EXE-346 on the mPDAI endoscopic subscore from baseline to day 57.
Phase 2: Change in EPS | 8 weeks
  To evaluate the effect of EXE-346 on EPS after 8 weeks.
Phase 2: Change in Fecal Calprotectin Level | 8 weeks
  To evaluate the effect of EXE-346 on fecal calprotectin levels after 8 weeks. The change from baseline fecal calprotectin level will be evaluated at Day 15, Day 29, and Day 57.
Phase 2: Change in SF-36 Score | 8 weeks
  To evaluate the effect of EXE-346 on patient reported outcomes after 8 weeks. Change in 36 items Short Form Survey Instrument (SF-36) score from baseline will be calculated at Day 29 and Day 57.
Phase 2: Change in GI PROMIS Score | 8 weeks
  To evaluate the effect of EXE-346 on patient reported outcomes after 8 weeks. Change in Gastrointestinal Patient Reported Outcomes Measurement Information System (GI PROMIS) score from baseline will be calculated at Day 29 and Day 57.
Phase 2: Percentage of Subjects Initiating Prohibited Medications | 8 weeks
  To assess the effect of EXE-346 on use of prohibited medications. Percentage of subjects who have initiated prohibited medication will be calculated at each study visit.
Phase 2 Open Label: Bowel Movement Frequency | 8 weeks
  To assess the effect of EXE-346 on bowel movement frequency using change in average daily bowel movement frequency from baseline and open-label baseline (baseline-OL) to each post-baseline week.
Phase 2 Open Label: Nighttime Awakening Frequency | 8 weeks
  To assess the effect of EXE-346 on nighttime awakening frequency using change in average nighttime awakening frequency from baseline and open-label baseline (baseline-OL) to each post-baseline week.
Phase 2 Open Label: Bowel Movement Consistency | 8 weeks
  To assess the effect of EXE-346 on bowel movement consistency using change in average consistency of daily bowel movements from baseline and open-label baseline (baseline-OL) to each post-baseline week
Phase 2 Open Label: Change in mPDAI Clinical Subscores | 8 weeks
  To evaluate the effect of EXE-346 on the mPDAI clinical subscores after 8 weeks. Change in clinical subscores will be from baseline and open-label baseline (baseline-OL) to each post-baseline visit.
Phase 2 Open Label: Change in Fecal Calprotectin | 8 weeks
  To evaluate the effect of EXE-346 on fecal calprotectin levels. The change in fecal calprotectin will be calculated from baseline and open-label baseline (baseline-OL) to each post-baseline visit.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Collins, MS, Study Director — Exegi Pharma, LLC
Locations (8):
- United States (8):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mayo Clinic - Florida (Inflammatory Bowel Disease Center), Jacksonville, Florida
  - Corewell Health, Grand Rapids, Michigan
  - Mayo Clinic Department of Gastroenterology, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Penn State Health (Milton S. Hershey Medical Center), Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allison J, Herrinton LJ, Liu L, Yu J, Lowder J. Natural history of severe ulcerative colitis in a community-based health plan. Clin Gastroenterol Hepatol. 2008 Sep;6(9):999-1003. doi: 10.1016/j.cgh.2008.05.022. PMID 18774533
- [Background] Barnes EL, Herfarth HH, Sandler RS, Chen W, Jaeger E, Nguyen VM, Robb AR, Kappelman MD, Martin CF, Long MD. Pouch-Related Symptoms and Quality of Life in Patients with Ileal Pouch-Anal Anastomosis. Inflamm Bowel Dis. 2017 Jul;23(7):1218-1224. doi: 10.1097/MIB.0000000000001119. PMID 28426474
- [Background] Biancone L, Michetti P, Travis S, Escher JC, Moser G, Forbes A, Hoffmann JC, Dignass A, Gionchetti P, Jantschek G, Kiesslich R, Kolacek S, Mitchell R, Panes J, Soderholm J, Vucelic B, Stange E; European Crohn's and Colitis Organisation (ECCO). European evidence-based Consensus on the management of ulcerative colitis: Special situations. J Crohns Colitis. 2008 Mar;2(1):63-92. doi: 10.1016/j.crohns.2007.12.001. Epub 2008 Jan 28. No abstract available. PMID 21172196
- [Background] Bibiloni R, Fedorak RN, Tannock GW, Madsen KL, Gionchetti P, Campieri M, De Simone C, Sartor RB. VSL#3 probiotic-mixture induces remission in patients with active ulcerative colitis. Am J Gastroenterol. 2005 Jul;100(7):1539-46. doi: 10.1111/j.1572-0241.2005.41794.x. PMID 15984978
- [Background] Bischoff SC, Escher J, Hebuterne X, Klek S, Krznaric Z, Schneider S, Shamir R, Stardelova K, Wierdsma N, Wiskin AE, Forbes A. ESPEN practical guideline: Clinical Nutrition in inflammatory bowel disease. Clin Nutr. 2020 Mar;39(3):632-653. doi: 10.1016/j.clnu.2019.11.002. Epub 2020 Jan 13. PMID 32029281
- [Background] Devaraj B, Kaiser AM. Surgical management of ulcerative colitis in the era of biologicals. Inflamm Bowel Dis. 2015 Jan;21(1):208-20. doi: 10.1097/MIB.0000000000000178. PMID 25222665
- [Background] Farouk R, Pemberton JH, Wolff BG, Dozois RR, Browning S, Larson D. Functional outcomes after ileal pouch-anal anastomosis for chronic ulcerative colitis. Ann Surg. 2000 Jun;231(6):919-26. doi: 10.1097/00000658-200006000-00017. PMID 10816636
- [Background] Gionchetti P, Calafiore A, Riso D, Liguori G, Calabrese C, Vitali G, Laureti S, Poggioli G, Campieri M, Rizzello F. The role of antibiotics and probiotics in pouchitis. Ann Gastroenterol. 2012;25(2):100-105. PMID 24714229
- [Background] Gionchetti P, Rizzello F, Helwig U, Venturi A, Lammers KM, Brigidi P, Vitali B, Poggioli G, Miglioli M, Campieri M. Prophylaxis of pouchitis onset with probiotic therapy: a double-blind, placebo-controlled trial. Gastroenterology. 2003 May;124(5):1202-9. doi: 10.1016/s0016-5085(03)00171-9. PMID 12730861
- [Background] Gionchetti P, Rizzello F, Morselli C, Poggioli G, Tambasco R, Calabrese C, Brigidi P, Vitali B, Straforini G, Campieri M. High-dose probiotics for the treatment of active pouchitis. Dis Colon Rectum. 2007 Dec;50(12):2075-82; discussion 2082-4. doi: 10.1007/s10350-007-9068-4. Epub 2007 Oct 13. PMID 17934776
- [Background] Gionchetti P, Rizzello F, Venturi A, Brigidi P, Matteuzzi D, Bazzocchi G, Poggioli G, Miglioli M, Campieri M. Oral bacteriotherapy as maintenance treatment in patients with chronic pouchitis: a double-blind, placebo-controlled trial. Gastroenterology. 2000 Aug;119(2):305-9. doi: 10.1053/gast.2000.9370. PMID 10930365
- [Background] Gower-Rousseau C, Dauchet L, Vernier-Massouille G, Tilloy E, Brazier F, Merle V, Dupas JL, Savoye G, Balde M, Marti R, Lerebours E, Cortot A, Salomez JL, Turck D, Colombel JF. The natural history of pediatric ulcerative colitis: a population-based cohort study. Am J Gastroenterol. 2009 Aug;104(8):2080-8. doi: 10.1038/ajg.2009.177. Epub 2009 May 12. PMID 19436273
- [Background] Hahnloser D, Pemberton JH, Wolff BG, Larson DR, Crownhart BS, Dozois RR. Results at up to 20 years after ileal pouch-anal anastomosis for chronic ulcerative colitis. Br J Surg. 2007 Mar;94(3):333-40. doi: 10.1002/bjs.5464. PMID 17225210
- [Background] Herrinton LJ, Liu L, Lewis JD, Griffin PM, Allison J. Incidence and prevalence of inflammatory bowel disease in a Northern California managed care organization, 1996-2002. Am J Gastroenterol. 2008 Aug;103(8):1998-2006. doi: 10.1111/j.1572-0241.2008.01960.x. PMID 18796097
- [Background] Hoffmann JC, Zeitz M, Bischoff SC, Brambs HJ, Bruch HP, Buhr HJ, Dignass A, Fischer I, Fleig W, Folsch UR, Herrlinger K, Hohne W, Jantschek G, Kaltz B, Keller KM, Knebel U, Kroesen AJ, Kruis W, Matthes H, Moser G, Mundt S, Pox C, Reinshagen M, Reissmann A, Riemann J, Rogler G, Schmiegel W, Scholmerich J, Schreiber S, Schwandner O, Selbmann HK, Stange EF, Utzig M, Wittekind C. [Diagnosis and therapy of ulcerative colitis: results of an evidence based consensus conference by the German society of Digestive and Metabolic Diseases and the competence network on inflammatory bowel disease]. Z Gastroenterol. 2004 Sep;42(9):979-83. doi: 10.1055/s-2004-813510. No abstract available. German. PMID 15455267
- [Background] Hurst RD, Molinari M, Chung TP, Rubin M, Michelassi F. Prospective study of the incidence, timing and treatment of pouchitis in 104 consecutive patients after restorative proctocolectomy. Arch Surg. 1996 May;131(5):497-500; discussion 501-2. doi: 10.1001/archsurg.1996.01430170043007. PMID 8624195
- [Background] Kappelman MD, Rifas-Shiman SL, Kleinman K, Ollendorf D, Bousvaros A, Grand RJ, Finkelstein JA. The prevalence and geographic distribution of Crohn's disease and ulcerative colitis in the United States. Clin Gastroenterol Hepatol. 2007 Dec;5(12):1424-9. doi: 10.1016/j.cgh.2007.07.012. Epub 2007 Sep 29. PMID 17904915
- [Background] Kmiot WA, Hesslewood SR, Smith N, Thompson H, Harding LK, Keighley MR. Evaluation of the inflammatory infiltrate in pouchitis with 111In-labeled granulocytes. Gastroenterology. 1993 Apr;104(4):981-8. doi: 10.1016/0016-5085(93)90264-d. PMID 8462824
- [Background] Langholz E, Munkholm P, Davidsen M, Binder V. Course of ulcerative colitis: analysis of changes in disease activity over years. Gastroenterology. 1994 Jul;107(1):3-11. doi: 10.1016/0016-5085(94)90054-x. PMID 8020674
- [Background] Loftus CG, Loftus EV Jr, Harmsen WS, Zinsmeister AR, Tremaine WJ, Melton LJ 3rd, Sandborn WJ. Update on the incidence and prevalence of Crohn's disease and ulcerative colitis in Olmsted County, Minnesota, 1940-2000. Inflamm Bowel Dis. 2007 Mar;13(3):254-61. doi: 10.1002/ibd.20029. PMID 17206702
- [Background] Madiba TE, Bartolo DC. Pouchitis following restorative proctocolectomy for ulcerative colitis: incidence and therapeutic outcome. J R Coll Surg Edinb. 2001 Dec;46(6):334-7. PMID 11768572
- [Background] Michelassi F, Lee J, Rubin M, Fichera A, Kasza K, Karrison T, Hurst RD. Long-term functional results after ileal pouch anal restorative proctocolectomy for ulcerative colitis: a prospective observational study. Ann Surg. 2003 Sep;238(3):433-41; discussion 442-5. doi: 10.1097/01.sla.0000086658.60555.ea. PMID 14501509
- [Background] Mimura T, Rizzello F, Helwig U, Poggioli G, Schreiber S, Talbot IC, Nicholls RJ, Gionchetti P, Campieri M, Kamm MA. Once daily high dose probiotic therapy (VSL#3) for maintaining remission in recurrent or refractory pouchitis. Gut. 2004 Jan;53(1):108-14. doi: 10.1136/gut.53.1.108. PMID 14684584
- [Background] Mowat C, Cole A, Windsor A, Ahmad T, Arnott I, Driscoll R, Mitton S, Orchard T, Rutter M, Younge L, Lees C, Ho GT, Satsangi J, Bloom S; IBD Section of the British Society of Gastroenterology. Guidelines for the management of inflammatory bowel disease in adults. Gut. 2011 May;60(5):571-607. doi: 10.1136/gut.2010.224154. PMID 21464096
- [Background] Ng SC, Plamondon S, Kamm MA, Hart AL, Al-Hassi HO, Guenther T, Stagg AJ, Knight SC. Immunosuppressive effects via human intestinal dendritic cells of probiotic bacteria and steroids in the treatment of acute ulcerative colitis. Inflamm Bowel Dis. 2010 Aug;16(8):1286-98. doi: 10.1002/ibd.21222. PMID 20155842
- [Background] Nguyen N, Zhang B, Holubar SD, Pardi DS, Singh S. Treatment and prevention of pouchitis after ileal pouch-anal anastomosis for chronic ulcerative colitis. Cochrane Database Syst Rev. 2019 Nov 30;11(11):CD001176. doi: 10.1002/14651858.CD001176.pub5. PMID 31785173
- [Background] Pardi DS, D'Haens G, Shen B, Campbell S, Gionchetti P. Clinical guidelines for the management of pouchitis. Inflamm Bowel Dis. 2009 Sep;15(9):1424-31. doi: 10.1002/ibd.21039. PMID 19685489
- [Background] Pathirana WGW, Chubb SP, Gillett MJ, Vasikaran SD. Faecal Calprotectin. Clin Biochem Rev. 2018 Aug;39(3):77-90. PMID 30828114
- [Background] Pronio A, Montesani C, Butteroni C, Vecchione S, Mumolo G, Vestri A, Vitolo D, Boirivant M. Probiotic administration in patients with ileal pouch-anal anastomosis for ulcerative colitis is associated with expansion of mucosal regulatory cells. Inflamm Bowel Dis. 2008 May;14(5):662-8. doi: 10.1002/ibd.20369. PMID 18240282
- [Background] Sagar PM, Taylor BA, Godwin P, Holdsworth PJ, Johnston D, Lewis W, Miller A, Quirke P, Williamson M. Acute pouchitis and deficiencies of fuel. Dis Colon Rectum. 1995 May;38(5):488-93. doi: 10.1007/BF02148848. PMID 7736879
- [Background] Sedano R, Ma C, Pai RK, D' Haens G, Guizzetti L, Shackelton LM, Remillard J, Gionchetti P, Gordon IO, Holubar S, Kayal M, Lauwers GY, Pai RK, Pardi DS, Samaan MA, Schaeffer DF, Shen B, Silverberg MS, Feagan BG, Sandborn WJ, Jairath V. An expert consensus to standardise clinical, endoscopic and histologic items and inclusion and outcome criteria for evaluation of pouchitis disease activity in clinical trials. Aliment Pharmacol Ther. 2021 May;53(10):1108-1117. doi: 10.1111/apt.16328. Epub 2021 Mar 18. PMID 33735522
- [Background] Shen B. Acute and chronic pouchitis--pathogenesis, diagnosis and treatment. Nat Rev Gastroenterol Hepatol. 2012 Apr 17;9(6):323-33. doi: 10.1038/nrgastro.2012.58. PMID 22508158
- [Background] Shen B, Achkar JP, Connor JT, Ormsby AH, Remzi FH, Bevins CL, Brzezinski A, Bambrick ML, Fazio VW, Lashner BA. Modified pouchitis disease activity index: a simplified approach to the diagnosis of pouchitis. Dis Colon Rectum. 2003 Jun;46(6):748-53. doi: 10.1007/s10350-004-6652-8. PMID 12794576
- [Background] Shen B, Achkar JP, Lashner BA, Ormsby AH, Remzi FH, Brzezinski A, Bevins CL, Bambrick ML, Seidner DL, Fazio VW. A randomized clinical trial of ciprofloxacin and metronidazole to treat acute pouchitis. Inflamm Bowel Dis. 2001 Nov;7(4):301-5. doi: 10.1097/00054725-200111000-00004. PMID 11720319
- [Background] Singh S, Feuerstein JD, Binion DG, Tremaine WJ. AGA Technical Review on the Management of Mild-to-Moderate Ulcerative Colitis. Gastroenterology. 2019 Feb;156(3):769-808.e29. doi: 10.1053/j.gastro.2018.12.008. Epub 2018 Dec 18. PMID 30576642
- [Background] Sood A, Midha V, Makharia GK, Ahuja V, Singal D, Goswami P, Tandon RK. The probiotic preparation, VSL#3 induces remission in patients with mild-to-moderately active ulcerative colitis. Clin Gastroenterol Hepatol. 2009 Nov;7(11):1202-9, 1209.e1. doi: 10.1016/j.cgh.2009.07.016. Epub 2009 Jul 22. PMID 19631292
- [Background] Spiegel BM, Reid MW, Bolus R, Whitman CB, Talley J, Dea S, Shahedi K, Karsan H, Teal C, Melmed GY, Cohen E, Fuller G, Yen L, Hodgkins P, Erder MH. Development and validation of a disease-targeted quality of life instrument for chronic diverticular disease: the DV-QOL. Qual Life Res. 2015 Jan;24(1):163-79. doi: 10.1007/s11136-014-0753-1. Epub 2014 Jul 25. PMID 25059533
- [Background] Tursi A, Brandimarte G, Papa A, Giglio A, Elisei W, Giorgetti GM, Forti G, Morini S, Hassan C, Pistoia MA, Modeo ME, Rodino' S, D'Amico T, Sebkova L, Sacca' N, Di Giulio E, Luzza F, Imeneo M, Larussa T, Di Rosa S, Annese V, Danese S, Gasbarrini A. Treatment of relapsing mild-to-moderate ulcerative colitis with the probiotic VSL#3 as adjunctive to a standard pharmaceutical treatment: a double-blind, randomized, placebo-controlled study. Am J Gastroenterol. 2010 Oct;105(10):2218-27. doi: 10.1038/ajg.2010.218. Epub 2010 Jun 1. PMID 20517305
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914